CLINICAL TRIAL: NCT04053309
Title: Implementation of a Round Spermatid Injection Protocol in a Clinical Infertility Practice
Brief Title: Round Spermatid Injection Protocol
Acronym: ROSI
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2019-03
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Male Infertility Due to Azoospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a blood sample of buccal swab will be obtained for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Males undergoing TESE or microTESE: All male patients undergoing surgical sperm extraction (TESE or microTESE) procedures as part of an IVF cycle at our center will be reviewed for inclusion and offered participation in the study. These men have been previously consented to the TESE or microTESE procedure at our center. The study will utilize the otherwise discarded round spermatids found in the TESE and microTESE surgical samples as the study samples being used for the ROSI procedure.

SUMMARY:
To evaluate embryology outcomes after application of a technique known as round spermatid injection (ROSI) into donor oocytes in a high-volume clinical infertility practice.

DETAILED DESCRIPTION:
The objective of this study is to assess embryology outcomes after implementation of a laboratory protocol known as ROSI at a high-volume clinical infertility practice. All samples from enrolled male patients with azoospermia who proceed with surgical sperm extraction (TESE or microTESE) will be evaluated for the presence of round spermatids. These round spermatids will be used as research samples as opposed to being discarded.

The investigators aim to identify whether the injection of round spermatids into donor oocytes can lead to successful fertilization, progression to the blastocyst stage, and euploid status. Performance of ROSI using donor oocytes not intended for implantation will allow the investigators to gain valuable insight regarding fertilization and development without any direct risk to patients or future offspring. These embryos are being generated for research purposes only and will ultimately be destroyed after the study has concluded. The investigators will measure rates of isolation of round spermatids from surgical samples, fertilization rates using donor oocytes, rates of progression to the blastocyst stage, and rates of aneuploidy using the previously described technique of ROSI.

ELIGIBILITY:
Major Inclusion Criteria: The following are major inclusion criteria:

1. A diagnosis of azoospermia after semen analysis.
2. Indication to proceed with testicular sperm extraction (TESE or microTESE) based on a urologic evaluation.
3. Presence of round spermatids from testicular sperm extraction (TESE or microTESE), irrespective of the presence or absence of mature spermatozoa.

Major Exclusion Criteria (must not meet any): The following are exclusion criteria:

1. Under 18 years old
2. All patients who do not voluntarily give their written consent for participation.
3. Men who do not wish to use their gametes (round spermatids) for fertilization of donor oocytes for research purposes.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: At least 10 healthy oocyte donors and at least 10 male patients with a diagnosis of male factor infertility (undergoing TESE or microTESE) to participate in this study.
  All male patients undergoing surgical sperm extraction (TESE or microTESE) procedures as part of an IVF cycle at our center will be reviewed for inclusion and offered participation in the study. These men have been previously consented to the TESE or microTESE procedure at our center. The study will utilize the otherwise discarded round spermatids found in the TESE and microTESE surgical samples as the study samples being used for the ROSI procedure.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Euploid blastulation rate | 1-2 weeks
  number of fertilized eggs progressing to the blastocyst stage of development which are euploid

SECONDARY OUTCOMES:
Fertilization Rate | 1 day post intracytoplasmic sperm injection procedure
  Number of mature eggs fertilized by round spermatids
Prevalence of round spermatids in surgical sperm samples | immediately after the TESE or microTESE
  the number of round spermatids present after a TESE or microTESE procedure is performed
Overall blastulation rate | 1 week
  number of fertilized eggs progressing to the blastocyst stage of development
Aneuploidy rate | 2 weeks
  the number of abnormal embryos after PGT-A

CONTACTS AND LOCATIONS:
Overall Officials: Brent Hanson, MD, Study Director — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No